CLINICAL TRIAL: NCT01891955
Title: Alimentation and Diabetes in Lanzarote - ADILAN: a Randomized Cross-over Pilot Trial Comparing a Healthy Diet With Grains and Dairy to a Healthy Diet Without Grains and Dairy in Patients With Type 2 Diabetes
Brief Title: Alimentation and Diabetes in Lanzarote - ADILAN: a Pilot Trial
Acronym: ADILAN
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Lund University (Other)
Collaborators: Cabildo de Lanzarote (Unknown); Ayuntamiento de Teguise (Unknown); Ayuntamiento de Arrecife (Unknown)
Responsible Party: Principal Investigator, Maelán Fontes-Villalba, PhD Student, Lund University
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: MFV-ADI-2013-01
Record Dates: First submitted 2013-06-28; First posted 2013-07-03 (Estimated); Last update posted 2014-03-21 (Estimated); Status verified 2014-03

CONDITIONS: Type 2 Diabetes
Keywords: Diabetes mellitus type 2; Cereals; Dairy; Dietary carbohydrates; Dietary fiber; Food; Metabolic syndrome; Satiety
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Metabolic Syndrome

ARMS (2):
- Diet A (Active Comparator): Healthy diet with grains and dairy
  Interventions: Behavioral: Healthy diet A
- Diet B (Active Comparator): Healthy diet without grains and dairy
  Interventions: Behavioral: Healthy diet B

INTERVENTIONS:
Behavioral: Healthy diet A — Healthy diet A will include fruit, vegetables, fish, shellfish, lean meat, nuts, eggs and olive oil. Macro/micronutrient composition, fiber intake and glycemic load will not differ from healthy diet B. Healthy diet A will include substantial amounts of whole grains, low-fat dairy and legumes (this is called "healthy diet with grains and dairy"). This diet is classified as very healthy using validated nutritional software. It is in accordance with official Spanish dietary recommendations for people with diabetes type 2 regarding macronutrient composition, dietary fiber, minerals and vitamins.
  Arms: Diet A
Behavioral: Healthy diet B — Healthy diet B will include fruit, vegetables, fish, shellfish, lean meat, nuts, eggs and olive oil. Macro/micronutrient composition, fiber intake and glycemic load will not differ from healthy diet A. Healthy diet B will exclude grains, legumes and dairy, which will largely be replaced by root vegetables, vegetables and fruit, and slightly more lean meat, fish and nuts (this is called "healthy diet without grains and dairy"). Salt intake will be lower in healthy diet B. This diet is classified as very healthy using validated nutritional software. It is in accordance with official Spanish dietary recommendations for people with diabetes type 2 regarding macronutrient composition, dietary fiber, minerals and vitamins.
  Arms: Diet B

SUMMARY:
The purpose of this study is to compare two healthy diets (according to official Spanish guidelines) that have been shown to be effective in the treatment of type 2 diabetes in order to see if one is better than the other.

Another goal is to test the hypothesis that food choice has metabolic effects that are independent of macro/micronutrient composition, fiber content, glycemic load and weight loss in the treatment of type 2 diabetes.

DETAILED DESCRIPTION:
There is some uncertainty with respect to the optimal dietary treatment of type 2 diabetes. In addition to energy balance, macronutrient composition, dietary fiber and glycemic load, increasing evidence suggests that the direct endocrine effects of food may be important.

In this trial, the intervention is based on two diets. The healthy diet with grains and dairy is based on whole grains, low-fat dairy, fish, shellfish, fruit, vegetables, legumes, eggs, nuts and refined vegetable oils rich in monounsaturated fatty acids (this is called "healthy diet A"). The healthy diet without grains and dairy is based on fish, shellfish, lean meat, fruit, vegetables, root vegetables, eggs and nuts, but excludes grains, legumes, refined vegetable oils, dairy products and salt (this is called "healthy diet B"). Both diets were classified as very healthy using validated nutritional software, and are considered healthy regarding macronutrient composition, fiber, mineral and vitamin intake according to the official Spanish dietary guidelines. The macro and micronutrient ratios, fiber content and glycemic load in healthy diet A and healthy diet B have been set to be equal.

The goal is to include 15 patients (>18 years) with medical diagnosis of type 2 diabetes, with or without medication, and increased waist circumference (≥80 cm for women and ≥94 cm for men), to a cross-over trial during two periods of 4-weeks separated by a 6-week washout period.

Lunch will be served in a hospital kitchen for control of nutrient intake, while the rest of meals will be eaten at home according to specific directions.

The working hypothesis of this study is that food choice has beneficial effects on the control of glucose beyond macro/micronutrient composition, fiber content, glycemic load and weight loss.

This study will provide information on whether food choice and diet quality has greater impact than macro/micronutrient composition, fiber content, glycemic load and weight loss in glucose control in patients with type 2 diabetes, and the need to conduct a long-term trial testing our hypothesis.

ELIGIBILITY:
Inclusion Criteria:

* Medical diagnosis of type 2 diabetes
* Increased waist circumference (≥80 cm for women and ≥94 cm for men)
* Unaltered medical diabetes treatment since three months before start of study
* Stable weight (varied less than 5%) since three months before start of study
* HbA1c ≥6.0%

Exclusion Criteria:

* Creatinine >130 μmol/L
* Change of treatment with betablocker last 3 months
* Change of treatment with thyroid hormone substitution last 3 months
* Treatment with anticoagulant medication
* Oral or injected steroid treatment
* Elevated liver enzymes (AST, ALT, ALP, GPT > 4 times their respective upper reference value)
* Physical or psychical illness, or changes in personal circumstances that make it impossible for the patient to continue in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2013-11; Primary Completion 2014-02 (Actual); Study Completion 2014-02 (Actual)

PRIMARY OUTCOMES:
Fasting fructosamine | Laboratory tests will be performed at baseline and after 4, 10 and 14 weeks
Fasting glucagon | Laboratory tests will be performed at baseline and after 4, 10 and 14 weeks

SECONDARY OUTCOMES:
Area under the curve for glucose (AUC glucose0-120) at the oral glucose tolerance test | Laboratory tests will be performed at baseline and after 4, 10 and 14 weeks
Area under the curve for glucagon (AUC glucagon0-120) at the oral glucose tolerance test | Laboratory tests will be performed at baseline and after 4, 10 and 14 weeks
Fasting plasma glucose | Laboratory tests will be performed at baseline and after 4, 10 and 14 weeks
Total cholesterol | Laboratory tests will be performed at baseline and after 4, 10 and 14 weeks
Low-density lipoprotein (LDL) cholesterol | Laboratory tests will be performed at baseline and after 4, 10 and 14 weeks
High-density lipoprotein (HDL) cholesterol | Laboratory tests will be performed at baseline and after 4, 10 and 14 weeks
Triglycerides | Laboratory tests will be performed at baseline and after 4, 10 and 14 weeks
Systolic and diastolic blood pressure | To be assessed at baseline and after 4, 10 and 14 weeks
High-sensitive C-reactive protein | Laboratory tests will be performed at baseline and after 4, 10 and 14 weeks
Waist circumference | To be assessed at baseline and after 4, 10 and 14 weeks
Hip circumference | To be assessed at baseline and after 4, 10 and 14 weeks
Sagittal abdominal diameter | To be assessed at baseline and after 4, 10 and 14 weeks
Tricipital, bicipital, suprailiac and subscapular skinfold thickness | To be assessed at baseline and after 4, 10 and 14 weeks
Satiation measured on a likert scale at food intake during 4 consecutive days | To be assessed at baseline and after 4, 10 and 14 weeks
Quality of life using a validated spanish version of the SF-36 questionnaire | To be assessed at baseline and after 4, 10 and 14 weeks
Change in medication | To be assessed at baseline and after 4, 10 and 14 weeks
Body weight | To be assessed at baseline and after 4, 10 and 14 weeks
Fasting HbA1c | Laboratory tests will be performed at baseline and after 4, 10 and 14 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Insular de Lanzarote, Arrecife, Las Palmas, Spain

REFERENCES:
- [Background] Nield L, Moore HJ, Hooper L, Cruickshank JK, Vyas A, Whittaker V, Summerbell CD. Dietary advice for treatment of type 2 diabetes mellitus in adults. Cochrane Database Syst Rev. 2007 Jul 18;2007(3):CD004097. doi: 10.1002/14651858.CD004097.pub4. PMID 17636747
- [Background] Ajala O, English P, Pinkney J. Systematic review and meta-analysis of different dietary approaches to the management of type 2 diabetes. Am J Clin Nutr. 2013 Mar;97(3):505-16. doi: 10.3945/ajcn.112.042457. Epub 2013 Jan 30. PMID 23364002
- [Background] Jonsson T, Granfeldt Y, Ahren B, Branell UC, Palsson G, Hansson A, Soderstrom M, Lindeberg S. Beneficial effects of a Paleolithic diet on cardiovascular risk factors in type 2 diabetes: a randomized cross-over pilot study. Cardiovasc Diabetol. 2009 Jul 16;8:35. doi: 10.1186/1475-2840-8-35. PMID 19604407
- [Background] Lindeberg S, Jonsson T, Granfeldt Y, Borgstrand E, Soffman J, Sjostrom K, Ahren B. A Palaeolithic diet improves glucose tolerance more than a Mediterranean-like diet in individuals with ischaemic heart disease. Diabetologia. 2007 Sep;50(9):1795-1807. doi: 10.1007/s00125-007-0716-y. Epub 2007 Jun 22. PMID 17583796
- [Background] Jonsson T, Olsson S, Ahren B, Bog-Hansen TC, Dole A, Lindeberg S. Agrarian diet and diseases of affluence--do evolutionary novel dietary lectins cause leptin resistance? BMC Endocr Disord. 2005 Dec 10;5:10. doi: 10.1186/1472-6823-5-10. PMID 16336696
- [Derived] Fontes-Villalba M, Jonsson T, Granfeldt Y, Frassetto LA, Sundquist J, Sundquist K, Carrera-Bastos P, Fika-Hernando M, Picazo O, Lindeberg S. A healthy diet with and without cereal grains and dairy products in patients with type 2 diabetes: study protocol for a random-order cross-over pilot study--Alimentation and Diabetes in Lanzarote--ADILAN. Trials. 2014 Jan 2;15:2. doi: 10.1186/1745-6215-15-2. PMID 24383431